CLINICAL TRIAL: NCT06132269
Title: Evaluation the Effect of AKK Formula on Intestinal Microbiota Regulation and Body Composition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: N202310027
Record Dates: First submitted 2023-11-09; First posted 2023-11-15 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Body Weight Changes; Metabolic Syndrome
Keywords: Akkermansia muciniphila
MeSH Terms: conditions — Body Weight Changes; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo sachet (Placebo Comparator): consume 1 sachet per day for 8 weeks
  Interventions: Dietary Supplement: Placebo sachet
- AKK formula sachet (Experimental): consume 1 sachet per day for 8 weeks
  Interventions: Dietary Supplement: AKK formula prebiotic sachet

INTERVENTIONS:
Dietary Supplement: AKK formula prebiotic sachet — 5 g/sachet, containing AKK formula, Indigestible Maltodextrin, Crystalline Maltitol, Calcium Carbonate, Citric Acid, Steviol Glycosides, and flavor.
  Subjects will consume 1 sachet per day for 8 weeks.
  Arms: AKK formula sachet
Dietary Supplement: Placebo sachet — 5 g/sachet, containing Indigestible Maltodextrin, Crystalline Maltitol, Calcium Carbonate, Citric Acid, Steviol Glycosides, and flavor.
  Subjects will consume 1 sachet per day for 8 weeks.
  Arms: Placebo sachet

SUMMARY:
The AKK formula, a prebiotic blend, can effectively promote the proliferation of A. muciniphila. In this study, we attempt to explore the clinical efficacy of AKK formula for A. muciniphila proliferation and weight management.

DETAILED DESCRIPTION:
This is a double-blind, randomized, parallel and placebo-controlled study. Subjects are informed to consume the samples daily for 8 weeks. The person who is evaluated as obesity by the investigator will be invited to participate in this trial. In this study, we attempt to explore the clinical efficacy of AKK formula for A. muciniphila proliferation and weight management.

ELIGIBILITY:
Inclusion Criteria:

* Subjects shall have a body mass index (BMI) of >23.0 to <32.5.0 kg/m2.
* Subjects shall have waist circumference of >80 cm for men and women.
* Subject is willing to maintain habitual dietary, lifestyle, and physical activity throughout the trial and do not plan to change the place of living during the study.
* Subject understands the study procedures and signs forms providing informed consent to participate in the study and authorizes the release of relevant protected health information to the Study Investigator.

Exclusion Criteria:

* Clinically important gastrointestinal condition that would potentially interfere with the evaluation of study products (e.g., inflammatory bowel disease, irritable bowel syndrome, gastric reflux, indigestion, dyspepsia, Crohn's disease, celiac disease, history of gastrointestinal surgical intervention for inducing weight loss, gastroparesis, and clinically significant lactose or gluten intolerance or other food/food component allergies).
* Recent (within 2 weeks of Visit 1, Day -7 - screening visit) history of an episode of acute GI illness such as nausea/vomiting or diarrhea (defined as >3 loose or liquid stools/d).
* Self-reported history (within 6 weeks of Visit 1, Day -7 -screening visit) of constipation (< 3 bowel movements/week) or diarrhea (loose stools >3 loose or liquid stools in one day) that in the judgement of the Study Investigator is not due to acute infection (e.g., stomach flu), food poisoning, temporary medication, etc.
* Subjests with mental disorder(depression, schizophrenia), cardiovascular disease/Arrhythmia/Heart Failure/Myocardial Infarction/or other Heart Condition, Hypothyroidism Or Uncontrolled Diabetic Gastrointestinal Disease (Crohn's Disease)/Gastrointestinal Resection Surgery/Irritable Bowel Syndrome, kidney condition, autoimmune disorder, Thyroid or hormonal abnormalities/Abnormalities If the immune system that can affect the weight of thyroid levels, like anemia/porphyrinosis, pancreatitis etc .
* Uncontrolled hypertension (systolic blood pressure ≥140 mm Hg or diastolic blood pressure ≥90 mm Hg) as defined by blood pressure measured on Visit 1. Stable use of hypertension medication is allowed (defined as no change in medication regimen within the 3 mo prior to Visit 1.)
* Any known food allergy, intolerance, or sensitivity to study product ingredients.
* Extreme dietary habits, eating disorders or physical activity patterns at the discretion of the Study Investigator.
* History or presence of cancer in the prior 2 years, except for non-melanoma skin cancer.
* Major trauma or any other surgical event within 3 months of Visit 1.
* Signs or symptoms of an active infection of clinical relevance within 5 days of Visit 1.
* Weight loss or gain >4.5 kg in the 3 months prior to Visit 1.
* Current use or planned use/participation in any weight loss regimen during the study period.
* Anti-biotic, antifungal, or antiparasitic use within 3 months of Visit 1 and throughout the study period.
* Use of anti-obesity, blood sugar lowering medications, insulin injections, hormones, diuretics , hormoneal treatment orsteroids within 1 month of Visit 1 and throughout the study period. Use of nasal and non-prescription topical treatments is permitted.
* Chronic use (i.e., daily or on a regular basis) of anti-inflammatory medications (e.g., NSAIDS) within 1 month of Visit 1.
* Use of medications (over-the-counter or prescription) and/or dietary supplements known to influence GI function including, but not limited to prebiotics, probiotics laxatives and/or enemas - including suppositories, fiber supplements, H2 blockers, proton pump inhibitors, antacids, anti-diarrheal agents, antidepressants, and/or anti-spasmodics within 3 weeks of Visit 1. Standard multi-vitamin/multi-mineral supplements are permitted.
* Subject has undergone endoscopy or endoscopy preparation within 3 months prior to Visit 1.
* Exposure to any non-registered drug product, including street drugs, within 4 weeks prior to Visit 1.
* Recent history (within 12 months of Visit 1) of alcohol or substance abuse. Alcohol abuse is defined as >14 drinks/week (1 drink = 12 oz (354 ml) beer, 5 oz (148 ml), or 1 ½ oz (44 ml) distilled spirits).
* Subject has a condition that, in the opinion of the Study Investigator, would interfere with his/her ability to provide informed consent, comply with the study protocol, confound interpretation of study results, or place the subject at undue risk.
* Female subjects who typically experience changes in GI symptoms or bowel habits (e.g., increased or decreased laxation, bloating, abdominal cramping) at the time of menstruation.
* Female subjects with irregular menstruation which does not allow for easy scheduling of stool collection outside of the menstrual period.
* Female subject who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period. Subjects who become pregnant during the study will be dismissed from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-11-09 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Relative abundance of Akkermansia muciniphila in gut | Change from Baseline relative abundance of A. muciniphila at 8 weeks
  Collect subject's feces for bacterial analysis. Akkermansia muciniphila will be quantified by quantitative PCR.
The change of waist circumference | Change from Baseline waist circumference at 4 weeks, and 8 weeks
  The waist circumference will be assessed by measuring tape. Unit: centimeter
The change of Waist-to-height ratio | Change from Baseline Waist-to-height at 4 weeks, and 8 weeks
  Waist-to-height ratio can be obtained by dividing waist size by height and is an effective indicator of risks associated with obesity.
The change of body mass index (BMI) | Change from Baseline BMI at 4 weeks, and 8 weeks
  BMI is a measurement of a person's leanness or corpulence based on their height and weight, and is intended to quantify tissue mass.The body mass index (BMI, kg/m^2) and body mass (kg) will be assessed by InBody.

SECONDARY OUTCOMES:
The change of total body mass | Change from Baseline total body mass at 4 weeks, and 8 weeks
  The total body mass (kg) will be assessed by Bioelectrical impedance analysis (BIA).
The change of total lean mass | Change from Baseline total lean mass at 4 weeks, and 8 weeks
  The total lean mass (kg) will be assessed by Bioelectrical impedance analysis (BIA).
The change of total fat mass | Change from Baseline total fat mass at 4 weeks, and 8 weeks
  The total fat mass (kg) will be assessed by Bioelectrical impedance analysis (BIA).
The change of total fat rate | Change from Baseline total fat rate at 4 weeks, and 8 weeks
  The total fat rate (%) will be assessed by Bioelectrical impedance analysis (BIA).
The change of visceral fat volume | Change from Baseline visceral fat volume at 4 weeks, and 8 weeks
  The visceral fat volume (cm^2) will be assessed by Bioelectrical impedance analysis (BIA).
The change of hip circumference | Change from Baseline hip circumference at 4 weeks, and 8 weeks
  The hip circumference will be assessed by measuring tape. Unit: centimeter
The change of insulin sensitivity | Change from Baseline insulin sensitivity at 8 weeks
  Insulin sensitivity is assessed by HOMA-IR. HOMA-IR= fasting insulin (microU/L) x fasting glucose (nmol/L)/22.5. Venous blood will be sampled to measure concentrations of fasting glycemia and insulin.
The change of total cholesterol | Change from Baseline total cholesterol at 8 weeks
  Venous blood will be sampled to measure concentrations of total cholesterol.
The change of High Density Lipoprotein Cholesterol (HDL-C) | Change from Baseline HDL-C at 8 weeks
  Venous blood will be sampled to measure concentrations of HDL-C.
The change of Low Density Lipoprotein Cholesterol (LDL-C) | Change from Baseline LDL-C at 8 weeks
  Venous blood will be sampled to measure concentrations of LDL-C.
The change of triglyceride | Change from Baseline triglyceride at 8 weeks
  Venous blood will be sampled to measure concentrations of triglyceride.
The change of intestinal microbiota | Change from Baseline intestinal microbiota at 8 weeks
  Collect subject's feces for bacterial analysis. Intestinal microbiota will be assessed by Next Generation Sequencing (NGS).
The change of gastrointestinal tolerability | Change from Baseline gastrointestinal tolerability at 4 weeks, and 8 weeks
  Gastointestinal tolerability will be assessed by The Gastrointestinal Symptom Rating Scale (GSRS).The GSRS has a seven-point graded Likert-type scale where 1 represents absence of troublesome symptoms and 7 represents very troublesome symptoms.
The change of stool type | Change from Baseline gastrointestinal tolerability at 4 weeks, and 8 weeks
  The stool type will be assessed by The Bristol Stool Form Scale (BSFS) daily. The BSFS is a scale that classifies stools, ranging from the hardest (type 1) to the softest (type 7).

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Ta Yang, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei, Taiwan